CLINICAL TRIAL: NCT02308059
Title: Diabetic Peripheral Neuropathy: Correlation Between Ultrasound Findings and Clinical Features
Brief Title: Ultrasonographic Evaluation of Diabetic Neuropathy
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Bayram Kelle, Director, Cukurova University
Other Study IDs: TF2012BAP13
Record Dates: First submitted 2014-12-01; First posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with diabetes mellitus: Group I; the patients with diabetes mellitus who had peripheral neuropathy as diagnosed.
  Interventions: Other: Ultrasonographic evaluation of nerves in diabetic patients
- Control: Group II; healthy volunteers
  Interventions: Other: Ultrasonographic evaluation of nerves of healthy volunteers

INTERVENTIONS:
Other: Ultrasonographic evaluation of nerves in diabetic patients — Ultrasonographic evaluation of peripheral nerves in patients with diabetes mellitus which have peripheral neuropathy
  Other Names: ultasonographic evaluation
  Groups: Patients with diabetes mellitus
Other: Ultrasonographic evaluation of nerves of healthy volunteers — evaluation of peripheral nerves and correlated with group I
  Groups: Control

SUMMARY:
The current study aimed to evaluate the cross-sectional area (CSA) of peripheral nerves in people with diabetic peripheral neuropathy using ultrasonography and correlate the CSA with clinical and demographic data.

DETAILED DESCRIPTION:
Patients with diabetic peripheral neuropathy (n=53) and a matched healthy control group (n=53) underwent blinded ultrasonography imaging of the sciatic, tibial and median nerves. Matching was performed according to patient body mass index (BMI), sex and age. CSAs of the nerves were recorded, and the associations between pain intensity (measured with a visual analog scale [VAS]), the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) pain scale, diabetes mellitus duration, BMI, HbA1c and blood glucose levels were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) scores ≥ 12
* probable diabetic peripheral neuropathy according to the diabetic peripheral neuropathy criteria.

Exclusion Criteria

* type 1 diabetes mellitus
* hypothyroidism
* LANSS pain scale scores < 12
* body mass index (BMI) > 35
* current pregnancy
* histories of hereditary neuropathy, inflammatory neuropathy, nerve trauma, or other known causes of polyneuropathy; and the use of anti-neuropathic drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients in a University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain scores on the visual analog scale | 3 years

SECONDARY OUTCOMES:
Neuropathic pain scores on the Leeds Assessment of Neuropathic Symptoms and Signs pain scale | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayram Kelle, Principal Investigator — Çukurova University, Faculty of Medicine